CLINICAL TRIAL: NCT01931267
Title: An Intervention Study of an Extended Discharge Planning and Disease Management Program on Patients With COPD
Brief Title: An Coach-based Intervention Study of an Extended Discharge Planning Program on Patients With COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 201112134RIC
Record Dates: First submitted 2013-06-10; First posted 2013-08-29 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Loss of Interest

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tablet Computer Motivated Instruction (Experimental): Using Tablet Computer Motivated Instruction to motivate patient learning breath skill and maintain practive. Research nurse will give 3 times instruction to patients during hospitalization. This arm estimated including 77 subjects.
  Interventions: Behavioral: Tablet Computer Motivated Instruction
- systematic instruction (Active Comparator): Research nurse give 3 times systematic instruction during hospitalization This arm estimated including 77 subjects.
  Interventions: Behavioral: Systematic Instruction

INTERVENTIONS:
Behavioral: Tablet Computer Motivated Instruction — Using tablet computer to motivate patient learning breath skill and maintain practive. Research nurse will give 3 times instruction to patients during hospitalization. This arm estimated including 77 subjects
  Arms: Tablet Computer Motivated Instruction
Behavioral: Systematic Instruction — Research nurse give 3 times systematic instruction during hospitalization This arm estimated including 77 subjects.
  Arms: systematic instruction

SUMMARY:
The purpose of this 4-year study is to investigate the relationship between cognition and learning ability on patients with COPD during hospitalization to establish and evaluate the effects of the community-extended discharge planning program. The transition theory is used as the theoretical base in this study. The patients with diagnosis of COPD in hospital will be invited to participate. The data of demographic variables, the cognitive function¸ the respiratory function, the effect of learning and the usage of medical resources after discharged will be collected. In the first year, we will establish the protocol of respiratory teaching in two modes, and to compare the differences among computer interaction game intervention, face to face teaching and routine nursing intervention, also to evaluate the related factors and the effect of learning on patients with COPD for determining the needs of patients' learning mode and the optimal frequency of nursing teaching mode during hospitalization in the second year. For the second year, build upon the results of the first year, the preliminary draft of the community-extended discharge planning program that base on the experts' meeting and the interview with the patients. Also, a pilot study that revising the content and testing the feasibility of respiratory teaching protocol will be conducted. For the 3rd and 4th year, using case-control RCT design, the community-extended discharge planning program will be tested in patients during their hospital stay and post-discharge period. The effects of this community-extended discharge planning program will be evaluated on outcome variables of patients' cognitive learning function, utilization of health care resources. The results of this study will help to develop a community-extended discharge planning for patients with COPD on cognition level and learning ability. Furthermore, the protocol of the community-extended discharge planning will serve as references to prolong the development of disease deterioration, reduce the probability of readmission and improve the quality of life.

DETAILED DESCRIPTION:
1. To establish the protocol of resiratory teaching mode.
2. To evaluate the related factors and the effect of learning on patients with COPD.
3. A modified discharge plan with respiratory teaching will implement to COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Being COPD Diagnosed Inpatients

Exclusion Criteria:

* Cancer with active treatment plan
* Lost speak ability
* Psychiatric problem
* Active TB

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
patient breath retraining skill | up to three months after discharge
  We held a professional commettee to draft a checklist(7 items) of breath retraining skill which comment to teach COPD patients. After retest and confirm the detail from pilot, we observated and rated patients breath retraing skill from none(0) to complete done(3). The higher points means the more correct skill that patients learned.

SECONDARY OUTCOMES:
self efficacy | baseline, one and three month after discharge
  PRAISAL questinnaire will be adopt after we consulted and get the author permission to use. Patients answered questionnaire(15 items) by their intuition. Rate point from 1 to 4 grades. The more confidence patient consider they have will rate more points. We propose patients learning the breath retraining skill well and correct during prepared discharge, they would get more confident.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Tzu Dai, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University, Taipai, Taiwan